CLINICAL TRIAL: NCT04853264
Title: ultraSound Guided PEripheral Catheterization Increases First-atTempt Success RAte in Hospitalized Patients When Compared With Conventional Technique: SPECTRA - Randomized Clinical Trial
Brief Title: Ultrasound Guided Peripheral Catheterization Increases First-attempt Success Rate
Acronym: SPECTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 39802620.0.0000.5327
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Venous Catheterization; Ultrasonography
Keywords: Peripheral venous catheterization; Ultrasonography; Nursing; Clinical trial; Randomized clinical trial

STUDY DESIGN:
Intervention Model Description: It's a randomized, parallel, controlled, blinded for data collection and analysis, single-center clinical trial; this study will follow the guidelines of the Consolidated Standards of Reporting Trials (CONSORT).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers and investigators responsible for data collection will be blinded for collection and analysis of data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: intervention group (Experimental): Ultrasound-guided peripheral venipuncture performed by a registered nurse with expertise in vascular access.
  Interventions: Device: Ultrasound-guided peripheral venipuncture
- Control group (Active Comparator): Conventional peripheral venipuncture performed by a registered nurse.
  Interventions: Device: Conventional peripheral venipuncture

INTERVENTIONS:
Device: Ultrasound-guided peripheral venipuncture — Ultrasound-guided peripheral venipuncture performed by a proficient vascular access registered nurse. The procedure will be performed according to the standard operational protocol for ultrasound guided peripheral venipuncture instituted at the hospital where the study will be conducted. Site Rite 8 or Site Rite 5 ultrasound machines (Bard Access Systems, Inc., USA) will be used on the procedures.
  Arms: Experimental: intervention group
Device: Conventional peripheral venipuncture — Conventional peripheral venipuncture performed by a registered nurse at the clinical inpatient unit. The procedure will be performed according to the standard operational protocol for peripheral venipuncture instituted in the hospital where the study will be conducted.
  Arms: Control group

SUMMARY:
Randomized clinical trial to test the assertiveness on the peripheral vein puncture attempt by comparing two methods: peripheral venipuncture catheterization using the conventional technique (vein visualization and palpation) versus ultrasound-guided venous puncture.

Patients with indication of peripheral venous puncture, admitted to the clinical inpatient units on the hospital where the study will be conducted (Hospital de Clinicas de Porto Alegre - HCPA) will be enrolled in this single-center trial and will be randomized to conventional peripheral venipuncture performed by a registered nurse; or ultrasound-guided peripheral venipuncture performed by a registered nurse with expertise in vascular access.

DETAILED DESCRIPTION:
Study Protocol:

When there is a need for peripheral venous access for the inpatient, the medical or nursing care team will contact the researchers, informing the personal data of the possible candidate to participate in the study. By fulfilling the eligibility criteria, the patient will be invited and informed about the study proposal; and, if he agrees to participate, he will sign the consent form. The type of procedure to be performed will be randomized through a draw. The procedure options are:

Intervention: peripheral venipuncture guided by ultrasound by a registered nurse with expertise in vascular access, or Control: conventional peripheral venipuncture by an inpatient care registered nurse.

Individuals who do not agree to participate in the study will have their data stored on a patient exclusion checklist.

In both groups, intervention and control, up to two attempts will be made by the same professional and, if there is no success on the procedure, another professional will be designated for two more attempts. Ultrasound Site Rite 8 or Ultrasound Site Rite 5, which are portable ultrasound devices that include 2D ultrasound imaging in real time, will be used on the Intervention Group (1) procedure.

The peripheral venipuncture procedure for both groups will be performed according to the standard operating procedures recommended by the institution where the study will be conducted (HCPA). The catheters to be used will be the peripheral venous catheters made available by the institution.

If there is a failure of puncture in the Control Group (2), the study participant will follow the institution's routine to adapt an appropriate vascular access, which is the activation of a nurse specialist in vascular access, who can perform peripheral venipuncture guided by ultrasound. In the event of a new insertion failure, the care team (doctor and nurse) discusses the case to define a new approach according to the infusional therapy, considering the protocol for the indication of venous vascular accesses at the institution. Thereafter, the patient can proceed for oral treatment, insertion of a peripherally inserted central catheter, insertion of a short-term central venous catheter, hypodermoclysis, long-term central venous catheter (totally or semi-implanted), according to the decision of the assistant team.

In the case of failure of the puncture in the Intervention Group (1), the study participant will follow the same routine of the institution, as explained above, for the adequacy of an adequate vascular access. However, in this case, the nurse specialist in vascular access will not be contacted, as the intervention procedure already uses ultrasound.

All participants who successfully insert a peripheral venous catheter in both groups will be monitored for the occurrence of any event related to the procedure from the time of insertion of the catheter until the loss of access for any reason, removal of the device at the end of therapy, discharge, death or eight days of follow-up, whichever comes first. Peripheral venous access that remains for more than eight days will be counted as event-free, access survival. Study participants with failed insertion will have the outcome computed in the database and will be followed up for another 48 hours to assess any complications resulting from the puncture attempt.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age = or > 18 years;
* Both sex;
* Admitted to the clinical inpatient units of the hospital where the study will be conducted (HCPA), with indication of peripheral venous puncture;
* Patients who do not configure emergency care.

Exclusion Criteria:

* Patients who have already received ultrasound-guided peripheral venipuncture at the current hospitalization;
* Patients in a critical or unstable clinical condition;
* Patients admitted to surgical units at HCPA;
* Patients in coronavirus (COVID-19) care units.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of venipuncture attempts | Immediately after the procedure.
  Success in the first attempt of venipuncture will be defined by the presence of blood reflux and infusion of 2 mL of saline without complaint of pain or signs of infiltration around the vessel.
  The number of times the vascular device reaches the skin and subcutaneous tissue with or without rupture of the vessel will be computed.

SECONDARY OUTCOMES:
Time to obtain peripheral venous access | During the procedure
  The time to obtain peripheral venous access will be measured in minutes. The computation of the total time of the procedure will start from the entry of the nurse into the patient's room and it will end when this professional leaves the room. In case of failure in venipuncture, the total time of the procedure will be considered as the sum of the time used in the procedure (without assertion) and the period necessary to obtain a functional venous access.
Classification of peripheral venous system conditions | Right before the procedure
  Predictors of difficult peripheral intravenous access will be recorded, considering demographic data (gender, age, weight, skin color, etc.) social behavior (active smoking, intravenous drug abuse and alcohol abuse), history of illnesses (heart and pulmonary diseases, vascular diseases, history of chemotherapy treatment, hematological status, use of drugs that interfere with cutaneous and vascular integrity, hypovolemia, hemodialysis, prolonged infusion therapies, skin changes, presence of scars and tattoos, dehydration, etc.) and history of difficult venous access.
Peripheral venous catheters characteristics | Before the procedure.
  Describe the technical specificities of the intravenous catheters used in the procedures, in terms of caliber and length.
Vascular and device complications | Up to 8 days.
  Complications that might occur during the permanence of the vascular access device (phlebitis, obstruction, leakage, infiltration, etc), measured through clinical assessment. In the case of the development of phlebitis, it will be evaluated through the application of the Visual Infusion Phlebitis Scale (from the Infusion Nurses Society), which classifies the lesion up to five degrees, according to the progression and severity of the signs and symptoms.
Venipuncture durability without complications | Up to 8 days.
  The time of permanence of the venous access without complications will be measured in days, counting from the day of insertion until the removal of the catheter for any reason (complications, end of therapy, discharge, death or eight days of follow-up). Venous accesses will follow the insertion site exchange guideline, that is, it will be exchange only when clinically indicated, in case of identified complication.
Infusional therapy characteristics and venipuncture durability | Up to 8 days.
  The characteristics of the prescribed intravenous therapy and the durability of peripheral venous access will be assessed daily using specific forms, developed by the authors. The following data will be collected regarding the prescribed intravenous therapy: medication in use, dose, frequency, and estimated duration of therapy.
Costs related to the venipuncture techniques used | Up to 8 days.
  Through specific forms, developed by the authors, the following will be computed: the number of catheters used, the complementary materials used and their quantities, the type of dressing for fixing the catheter and the time spent to obtain peripheral venous access.

CONTACTS AND LOCATIONS:
Overall Officials: Eneida R Rabelo-Silva, RN, MSc, ScD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Universidade Federal do Rio Grande do Sul - Post Graduated Program, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Database
Supporting Information: SAP, Analytic Code
Time Frame: After publication